CLINICAL TRIAL: NCT04129385
Title: Effect of Postoperative Trendelenburg Position on Shoulder Pain After Gynecological Laparoscopic Procedures.
Brief Title: Post Laparoscopy Shoulder Pain and Postoperative Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Nassif, Assistant Professor, Department of Obstetrics & Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AmericanUBMC1
Record Dates: First submitted 2019-06-28; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Shoulder Pain
Keywords: laparoscopy; shoulder pain; trendelenburg position
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group S (No Intervention): Control group (Group S: 54 patients); this group will undergo the standard laparoscopic procedure (the procedure is done in Trendelenburg position). While in Trendelenburg position and prior to wound closure and with laparoscopic port valves open, the patient's abdomen will be passively deflated. The patients will be placed in supine head up position in the post anesthesia care unit (PACU).
- Group T (Experimental): Intervention group (Group T: 54 patients); the patients will be subject to the same maneuver as in arm 1 prior to wound closure but will be positioned in a 20 degree Trendelenburg position once fully awake and cooperative in the PACU and will remain in this position for the first 24 hours post operatively, even after they are transferred to their rooms on the American University of Beirut Medical Center (AUBMC) floors. The maximum time allowed in a straight-up position will be three 15-minute intervals over a 24-hour period (the first interval being a clear fluids intake at 12 hours postoperatively).
  Interventions: Procedure: 20 degree Trendelenburg position

INTERVENTIONS:
Procedure: 20 degree Trendelenburg position — The patients in the intervention group will be placed in trendelenburg position postoperatively.
  Arms: Group T

SUMMARY:
Laparoscopic surgery has become a standard of care for many gynecological surgeries due to its lower morbidity, pain and cost compared to open techniques. Unfortunately, the use of carbon dioxide (CO2) to insufflate the abdomen is a major contributor to post operative shoulder pain. Shoulder pain post laparoscopy is common and it is a major cause of patient dissatisfaction. The aim of our study is to evaluate the efficacy of positioning the patient in Trendelenburg, post operatively for 24 hours, on shoulder pain reduction. Our hypothesis is based on the assumption that complete CO2 deflation is not possible and that Trendelenburg positioning will help displace CO2 from the sub diaphragmatic area thus reducing the diaphragmatic and phrenic nerve irritation causing pain.

DETAILED DESCRIPTION:
A prospective randomized controlled study with 54 patients in each of the two arms. Group S (control) will undergo the standard laparoscopic procedure and the patients will be placed in supine head up position postoperatively. In group T (interventional); the patients will be positioned in Trendelenburg position once fully awake and cooperative in the post-anesthesia case unit (PACU) and will remain in this position for the first 24 hours postoperatively. Postoperative NRS(numeric rating scale) score for shoulder pain and nausea will be collected at arrival to PACU, & 4, 6, 12 and 24 hours postoperatively. In addition, total amount of rescue pain and nausea medication used by the patient will be recorded. Data collected will be analyzed and compared between the two groups. The independent t- test will be used to compare postoperative shoulder pain, with NRS scores treated as continuous variable, between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age: 18 years to 60 years, American Society of Anesthesiologist physical status (ASA) 1 or 2
* Diagnostic or operative gynecologic laparoscopy {4 port sites, three 5 mm trocars (suprapubic, right and left iliac fossa) and one 10 mm trocar (umbilical)} between one and 3 hours duration.
* Abdominal incisions less than 1.5 cm.
* Steady abdominal insufflation pressure of 14 mm Hg following a gradual insufflation over a 5-minute period.
* Insufflation at a steady maximal flow of 30 l/min

Exclusion Criteria:

* Conversion to laparotomy.
* Abdominal insufflation pressure more than 14 mm Hg.
* Medical drug allergy to paracetamol, ketoprofen and/or tramadol.
* Presence of gastro-esophageal reflux (GERD)
* Pregnancy
* Patient with Thrombophilias and or at high risk of Deep Vein Thrombosis (DVT)
* Obesity body mass index (BMI) greater than 40
* One day surgery patients

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Shoulder pain (12 hours) | 12 hours after laparoscopic surgery
  Pain score (measured using a 0-10 numerical scale) at 12 hours

SECONDARY OUTCOMES:
Shoulder pain | at arrival to post anesthesia care unit (PACU), 4, 6, and 24 hours, after laparoscopic surgery
  Pain score (measured using a 0-10 numerical scale)
Presence of nausea | at arrival to PACU, 4, 6, 12 and 24 hours, after laparoscopic surgery
  Presence or absence of nausea (yes/no)
Severity of Nausea | at arrival to PACU, 4, 6, 12 and 24 hours, after laparoscopic surgery
  Nausea score (measured using a 0-10 numerical scale)
Rescue pain medication | within first 24 hours after laparoscopic surgery
  Time to first rescue pain medication (minutes)
Total rescue pain medication | within first 24 hours after laparoscopic surgery
  Total rescue pain medication during first 24 hours
Patient satisfaction | 24 hours post laparoscopic surgery
  Patient satisfaction with surgical experience (measured using a 0-10 numerical scale)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Nassif, M.D., Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett JC, Hurd WW, Rogers RM Jr, Williams NL, Shapiro SA. Laparoscopic positioning and nerve injuries. J Minim Invasive Gynecol. 2007 Sep-Oct;14(5):664-72; quiz 673. doi: 10.1016/j.jmig.2007.04.008. No abstract available. PMID 17848335
- [Background] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858
- [Background] Madsen MR, Jensen KE. Postoperative pain and nausea after laparoscopic cholecystectomy. Surg Laparosc Endosc. 1992 Dec;2(4):303-5. PMID 1341550
- [Background] Coventry DM. Anaesthesia for laparoscopic surgery. J R Coll Surg Edinb. 1995 Jun;40(3):151-60. PMID 7616466
- [Background] Korell M, Schmaus F, Strowitzki T, Schneeweiss SG, Hepp H. Pain intensity following laparoscopy. Surg Laparosc Endosc. 1996 Oct;6(5):375-9. PMID 8890423
- [Background] Jackson SA, Laurence AS, Hill JC. Does post-laparoscopy pain relate to residual carbon dioxide? Anaesthesia. 1996 May;51(5):485-7. doi: 10.1111/j.1365-2044.1996.tb07798.x. PMID 8694166
- [Background] Kojima Y, Yokota S, Ina H. Shoulder pain after gynaecological laparoscopy caused by arm abduction. Eur J Anaesthesiol. 2004 Jul;21(7):578-9. doi: 10.1017/s0265021504267126. No abstract available. PMID 15318475
- [Background] Lepner U, Goroshina J, Samarutel J. Postoperative pain relief after laparoscopic cholecystectomy: a randomised prospective double-blind clinical trial. Scand J Surg. 2003;92(2):121-4. PMID 12841551
- [Background] Berberoglu M, Dilek ON, Ercan F, Kati I, Ozmen M. The effect of CO2 insufflation rate on the postlaparoscopic shoulder pain. J Laparoendosc Adv Surg Tech A. 1998 Oct;8(5):273-7. doi: 10.1089/lap.1998.8.273. PMID 9820719
- [Background] Pergialiotis V, Vlachos DE, Kontzoglou K, Perrea D, Vlachos GD. Pulmonary recruitment maneuver to reduce pain after laparoscopy: a meta-analysis of randomized controlled trials. Surg Endosc. 2015 Aug;29(8):2101-8. doi: 10.1007/s00464-014-3934-7. Epub 2014 Nov 1. PMID 25361653
- [Background] Sharami SH, Sharami MB, Abdollahzadeh M, Keyvan A. Randomised clinical trial of the influence of pulmonary recruitment manoeuvre on reducing shoulder pain after laparoscopy. J Obstet Gynaecol. 2010;30(5):505-10. doi: 10.3109/01443611003802313. PMID 20604657
- [Background] Nezhat, C. and F. Nezhat, Nezhat's Operative Gynecologic Laparoscopy and Hysteroscopy2008: Cambridge University Press.
- [Background] Suginami R, Taniguchi F, Suginami H. Prevention of postlaparoscopic shoulder pain by forced evacuation of residual CO(2). JSLS. 2009 Jan-Mar;13(1):56-9. PMID 19366542
- [Derived] Zeeni C, Chamsy D, Khalil A, Abu Musa A, Al Hassanieh M, Shebbo F, Nassif J. Effect of postoperative Trendelenburg position on shoulder pain after gynecological laparoscopic procedures: a randomized clinical trial. BMC Anesthesiol. 2020 Jan 29;20(1):27. doi: 10.1186/s12871-020-0946-9. PMID 31996139